CLINICAL TRIAL: NCT06242262
Title: Deep Neuromuscular Block With Low Pressure Pneumoperitoneum in Laparoscopic Abdominal Surgeries: A Randomized Controlled Trial
Brief Title: Deep Neuromuscular Block With Low Pressure Pneumoperitoneum in Laparoscopic Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ِAhmed Mohamed Ibrahim, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR461/12/2023
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Deep Neuromuscular Block; Low Pressure; Pneumoperitoneum; Laparoscopic Abdominal Surgeries
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep neuromuscular block (Experimental): Patients will receive deep neuromuscular block by using cis-atracurium
  Interventions: Other: Deep neuromuscular block
- Moderate neuromuscular block (Other): Patients will receive moderate neuromuscular block by using cis-atracurium.
  Interventions: Other: Moderate neuromuscular block

INTERVENTIONS:
Other: Deep neuromuscular block — Patients will receive deep neuromuscular block by using cis-atracurium. After tracheal intubation for 15 min, a cis-atracurium pump will be started, and its rate will be adjusted to maintain a post-tetanic count (PTC) in the 1-2 range.
  Arms: Deep neuromuscular block
Other: Moderate neuromuscular block — Patients will receive moderate neuromuscular block by using cis-atracurium. Pump delivery of cis-atracurium will be started when the TOF count returned to 2. The TOF count is maintained between 1 and 3 by adjusting the pump rate
  Arms: Moderate neuromuscular block

SUMMARY:
The aim of this study is to evaluate the effect of deep neuromuscular block on postoperative pain, duration of surgery, quality of surgical field, length of recovery room stays, Total amount of rescue analgesic, postoperative nausea/vomiting, and length of hospital stay.

DETAILED DESCRIPTION:
Acute-pain management in surgery patients is accompanied by an array of negative consequences, including increased morbidity, impaired physical function, and quality of life, slowed recovery, prolonged opioid use during and after hospitalization, and increased cost of care.

Reducing pneumo-peritoneum (PP) is one technique for reducing postoperative pain. The effect of low PP on postoperative pain remains a controversial topic with other studies reporting no difference in postoperative pain levels between the Two pressures.

Deep neuromuscular block (DNMB) in abdominal surgeries is associated with various advantages, such as lower abdominal pressure, lower pain and rescue opioid consumption, as well as less bleeding. DNMB may facilitate the use of reduced insufflation pressure without compromising the surgical field of vision. However, its usage is limited due to a lack of predictable and rapid recovery with conventional NMB antagonists (neostigmine) or spontaneous recovery

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Patients scheduled for laparoscopic abdominal surgery.

Exclusion Criteria:

* Known allergies to cis-atracurium or neostigmine.
* Contraindications to the use of neostigmine, such as bronchial asthma, glaucoma, myocardial ischemia, and epilepsy.
* History of neuromuscular, renal, or hepatic disease; previous abdominal surgery.
* Treatment with drugs known to affect neuromuscular function.
* Preoperative hyperalgesia.
* Peripheral neuropathy is caused by diabetes.
* History of chronic analgesics treatment, drug, or alcohol abuse.
* Body mass index (BMI) > 35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain | 48 hours postoperatively
  The degree of pain will be evaluated using the numerical rating scale (NRS) from (0 to 10), zero means no pain and ten means the worst pain. It will be measured at PACU, 1h, 2h. 4hr, 6h, 8h, 12h, 18h, 24h, 36h and 48h postoperative.

SECONDARY OUTCOMES:
Time of first analgesic | 48 hours postoperatively
  Time of first analgesic will be measured from the end of surgery till first dose of morphine administrated. If numerical rating scale (NRS) is more than 3, intravenous morphine 3mg will be administered as rescue analgesia.
Total opioid consumption in 1st 48h | 48 hours postoperatively
  A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. If numerical rating scale (NRS) is more than 3, intravenous morphine 3mg will be administered as rescue analgesia.
The degree of Patient satisfaction | 48 hours postoperatively
  The degree of patient satisfaction will be assessed on a 5-point scale: (0= extremely dissatisfied, 1= unsatisfied, 2= neither satisfied nor unsatisfied, 3= satisfied), 4= extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.